CLINICAL TRIAL: NCT02121834
Title: A Multiple-Dose, Dose Escalation, Safety, Tolerability, and Pharmacokinetic Study of LY3050258
Brief Title: A Study of LY3050258 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14936; I6R-MC-DLAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY3050258 (Experimental): Daily dose of LY3050258 for 28 days: Cohort A 10 mg, Cohort B 30 mg, Cohort C 90 mg, Cohort D 180 mg and Cohort E 360 mg.
  Interventions: Drug: LY3050258; Drug: Placebo
- Placebo (Placebo Comparator): Daily dose of placebo matching LY3050258 for 28 days.
  Interventions: Drug: LY3050258; Drug: Placebo

INTERVENTIONS:
Drug: LY3050258
Drug: Placebo

SUMMARY:
This is a multiple dose study of LY3050258 in healthy men and postmenopausal women. This study will evaluate the safety and how well the body tolerates LY3050258. It will last approximately 14 weeks with a 2 week follow-up appointment after the last treatment with study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy postmenopausal females, including Japanese participants
* Body mass index (BMI) of 18 and 35 kilograms per square meter (kg/m^2), inclusive

Exclusion Criteria:

* Abnormal siting blood pressure as determined by the investigator
* Abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, places the participant at an unacceptable risk for study participation
* Aspartate aminotransferase (AST) or alkaline phosphatase (ALT) greater than 2 times the upper limit of normal (ULN)
* Skin condition that in the opinion of the investigator makes the participant unsuitable for study participation
* Current use of statins within the last 3 months prior to dosing
* Current use or previous use of anabolic steroids in the preceding 6 months prior to dosing
* Use of dehydroepiandrosterone, other potential over-the-counter steroidal supplements, or other nutritional products intended to have weight-reduction and/or performance-enhancing effects within 21 days prior to dosing

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A-D Placebo; Cohort E Placebo: Placebo daily for 28 days
- Cohort A: 10 Milligram (mg) LY3050258: 10 mg LY3050258, daily for 28 days
- Cohort B: 30 mg LY3050258: 30mg LY3050258, daily for 28 days
- Cohort C: 90 mg LY3050258: 90 mg LY3050258, daily for 28 days
- Cohort D: 180 mg LY3050258: 180 mg LY3050258, daily for 28 days
- Cohort E: 360 mg LY3050258: 360 mg LY3050258, daily for 28 days
Period: Overall Study
Arm/Group | Cohort A-D Placebo | Cohort A: 10 Milligram (mg) LY3050258 | Cohort B: 30 mg LY3050258 | Cohort C: 90 mg LY3050258 | Cohort D: 180 mg LY3050258 | Cohort E: 360 mg LY3050258 | Cohort E Placebo
Started | 12 | 11 | 9 | 10 | 9 | 9 | 3
Received at Least One Dose of Study Drug | 12 | 11 | 9 | 10 | 9 | 9 | 3
Completed | 12 | 9 | 7 | 10 | 9 | 9 | 3
Not Completed | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: LY3050258: 10 mg LY3050258, daily for 28 days
- Cohort B: LY3050258: 30 mg LY3050258, daily for 28 days
- Cohort C: LY3050258: 90 mg LY3050258, daily for 28 days
- Cohort D: LY3050258: 180 mg LY3050258, daily for 28 days
- Cohort E: LY3050258: 360 mg LY3050258, daily for 28 days
- Total: Total of all reporting groups
Arm/Group | Cohort A-D Placebo | Cohort A: LY3050258 | Cohort B: LY3050258 | Cohort C: LY3050258 | Cohort D: LY3050258 | Cohort E: LY3050258 | Cohort E Placebo | Total
Number analyzed (Participants) | 12 | 11 | 9 | 10 | 9 | 9 | 3 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (12.2) | 50.5 (9.8) | 51.6 (9.1) | 52.8 (10.4) | 44.6 (10.6) | 47.8 (10.5) | 35.7 (5.5) | 48.7 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 2 | 3 | 3 | 0 | 21
  Male | 8 | 5 | 6 | 8 | 6 | 6 | 3 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 2 | 3 | 0 | 5 | 2 | 17
  Not Hispanic or Latino | 12 | 6 | 7 | 7 | 9 | 4 | 1 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 2 | 3 | 3 | 2 | 1 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 1 | 4 | 1 | 0 | 14
  White | 6 | 5 | 5 | 6 | 2 | 5 | 2 | 31
  More than one race | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 9 | 10 | 9 | 9 | 3 | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: Clinically significant events were defined as serious and other nonserious adverse events (AE) related to study drug. A summary of other nonserious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline to Study Completion (Up to 14 Weeks)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Cohort A-D; Placebo Cohort E: Placebo daily for 28 days
- 10 mg LY3050258: 10 mg LY3050258, daily for 28 days
- 30 mg LY3050258: 30 mg LY3050258, daily for 28 days
- 90 mg LY3050258: 90 mg LY3050258, daily for 28 days
- 180 mg LY3050258: 180 mg LY3050258, daily for 28 days
- 360 mg LY3050258: 360 mg LY3050258, daily for 28 days
Arm/Group | Placebo Cohort A-D | 10 mg LY3050258 | 30 mg LY3050258 | 90 mg LY3050258 | 180 mg LY3050258 | 360 mg LY3050258 | Placebo Cohort E
Number analyzed (Participants) | 12 | 11 | 9 | 10 | 9 | 9 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve During One Dosing Interval at Steady State (AUC τ,ss) of Multiple Doses of LY3050258
Time Frame: Baseline through 4 weeks: Day 1 at 4,8,12, 18, and 24 hours (hrs); Day 7 at Pre-dose, 4,8,and 12 hrs; Day 14 at Pre-dose; Days 26 and 27 at Pre-dose; Day 28 at Pre-dose, 4, 8,12,18, and 24 hrs
Population: All participants who received at least one dose of study drug and had measurable AUC PK concentrations after dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- 10mg LY3050258: 10 mg LY3050258, daily for 28 days
- 30mg LY3050258: 30 mg LY3050258, daily for 28 days
- 90mg LY3050258: 90 mg LY3050258, daily for 28 days
- 180mg LY3050258: 180 mg LY3050258, daily for 28 days
- 360mg LY3050258: 360mg LY3050258, daily for 28 days
Arm/Group | 10mg LY3050258 | 30mg LY3050258 | 90mg LY3050258 | 180mg LY3050258 | 360mg LY3050258
Number analyzed (Participants) | 9 | 7 | 9 | 9 | 9
nanogram*hour per milliliter (ng*hr/mL) | 14.5 (81) | 24.1 (55) | 55.6 (62) | 70.0 (50) | 84.5 (65)

3. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Multiple Doses of LY3050258
Time Frame: as for outcome 2
Population: All participants who received at least one dose of study drug and had measurable Cmax PK concentrations after dosing.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 10 mg LY3050258 | 30 mg LY3050258 | 90 mg LY3050258 | 180 mg LY3050258 | 360 mg LY3050258
Number analyzed (Participants) | 9 | 8 | 9 | 9 | 9
nanogram per milliliter (ng/mL) | 0.899 (93) | 1.35 (63) | 3.58 (61) | 4.51 (57) | 4.99 (62)

ADVERSE EVENTS:
Groups:
- Cohort A: 10 mg LY3050258: 10 mg LY3050258, daily for 28 days
- Cohort B: 30 mg LY3050258: 30 mg LY3050258, daily for 28 days
- Cohort E: Placebo: Placebo daily for 28 days
Arm/Group | Cohort A-D Placebo | Cohort A: 10 mg LY3050258 | Cohort B: 30 mg LY3050258 | Cohort C: 90 mg LY3050258 | Cohort D: 180 mg LY3050258 | Cohort E: 360 mg LY3050258 | Cohort E: Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/9 | 0/10 | 0/9 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 5/12 | 4/11 | 2/9 | 3/10 | 6/9 | 4/9 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A-D Placebo (N=12) | Cohort A: 10 mg LY3050258 (N=11) | Cohort B: 30 mg LY3050258 (N=9) | Cohort C: 90 mg LY3050258 (N=10) | Cohort D: 180 mg LY3050258 (N=9) | Cohort E: 360 mg LY3050258 (N=9) | Cohort E: Placebo (N=3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Application site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other